CLINICAL TRIAL: NCT05574582
Title: Arthroscopic Versus Open Cancellous Bone Grafting for Scaphoid Delayed/Non-union in Adults: Study Protocol for a Randomized Clinical Trial
Brief Title: Arthroscopic vs. Open Bone Grafting for Scaphoid Delayed/Nonunion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Morten Kjaer, Medical doctor, PhD student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT Scaphoid delayed/nonunion
Record Dates: First submitted 2022-09-30; First posted 2022-10-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Scaphoid Fracture; Scaphoid Nonunion
Keywords: Scaphoid; Scaphoid nonunion; Cancellous; Graft; Arthroscopic; Timo to union
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: 1:1 observer-blinded randomized controlled, superiority trial. The main objective is to compare open C graft with arthroscopic assisted C chips graft reconstruction for scaphoid fractures with delayed/non-union.
  Based on the sample size calculation, a total of 88 patients with scaphoid delayed/non-union are randomized to either:
  1. Group A - Arthroscopic assisted C chips graft reconstruction (intervention group), n=44
  2. Group O - Open C graft reconstruction (control group), n=44
  The randomization is done in the outpatient clinic and the patients will be informed about the operative treatment. The randomization application, Research Electronic Data Capture (REDCap), will allocate patients in a 1:1 ratio, stratified for proximal pole fracture (yes /no), dislocation (>/< 2mm), and smoking (yes/ no). A statistician will generate a randomization sequence for REDCap.
Who Masked: Investigator, Outcomes Assessor
Masking Description: observer-blinded RCT, union is assessed by a blinded musculoskeletal radiologist. QDASH is a patient-reported survey, without the involvement of surgeons or research staff. Other secondary outcomes will be measured by an independent observer. The study will not be blinded to the operating theatre staff, surgeons, physiotherapists, or patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic assisted Cancellous chips graft reconstruction (Experimental): The arthroscopic technique is potentially less invasive with minimal donor site morbidity and potentially faster time to union because of minimal trauma to the ligament structures, joint capsule, and the tenuous blood supply. It may also have advantageous osteogenic properties compared to a structural graft.
  Currently, studies have reported similar union rates, patient reported outcomes score, and functional score compared to open graft technique. Results in patients with gross deformity are debated with some studies favoring conventional open structural graft and other found no difference in outcome between the techniques.
  Interventions: Procedure: Graft reconstruction and internal fixation with compression screw
- Open cancellous graft reconstruction (Active Comparator): Convention open technique with debridement of the nonunion side, insertion of cancellous graft from the iliac crest and osteosynthesis with compression screw is currently commonly applied in scaphoid nonunion.
  Interventions: Procedure: Graft reconstruction and internal fixation with compression screw

INTERVENTIONS:
Procedure: Graft reconstruction and internal fixation with compression screw — Patients suffering from scaphoid nonunion are treated surgically by debridement, graft reconstruction and internal fixation with compression screw

SUMMARY:
Single site, prospective, observer-blinded randomized controlled trial. Eighty-eight patients aged 18-68 years with scaphoid delayed/non-union, will be randomized, 1:1, to either open iliac crest cancellous graft reconstruction or arthroscopic assisted distal radius cancellous chips graft reconstruction. All Danish citizens, referred to the orthopedic department, Copenhagen University Hospital in Gentofte with scaphoid delayed/nonunion will be offered participation in the trial. Exclusion criteria are: Associated fracture in the hand/upper extremity, previous failed surgical treatment for scaphoid delayed/nonunion, stage 2 SNAC or above, avascular necrosis of the proximal pole and gross deformity.

Patients are stratified for smoking habits, proximal pole involvement, and displacement of >/<2mm. The primary outcome is time to union, measured with repeated CT scans at 2-week intervals from 6 to 16 weeks postoperatively. Secondary outcomes are Quick disabilities of the Arm, Shoulder and Hand (Q-DASH), Visual Analogue scale (VAS), donor site morbidity, union rate, restoration of scaphoid deformity, range of motion, key-pinch, grip strength, EQ5D-5L, patient satisfaction, complications, and revision surgery. Patients are examined before the operation and 1.5, 3, 6, 12 and 24 month after the operation. Online follow-up 5 and 10 years after surgery are performed.

DETAILED DESCRIPTION:
A scaphoid fracture is the most common injury to the carpal bones. The incidence is 107-151/100.000 per year and fractures are predominantly sustained by males in their twenties. Scaphoid non-union is defined as a lack of healing 6 months after injury and develops in 5-25% of cases after non-operative treatment. Delayed union is defined as incomplete healing 2-6 months after injury. However, some potential for a union probably exists, especially in nondisplaced fractures, otherwise this condition is associated with a transition into a persistent non-union. The risk of non-union increases with delayed diagnosis and treatment, displaced fractures, proximal pole fractures, smoking, poor vascularity, and advancing age.

The scaphoid is primarily covered with cartilage and has a retrograde blood supply. The dorsal branch of the radial artery accounts for 80% and a separate volar branch for 20 % of the extramedullary blood supply. The proximal pole is only supplied by the intramedullary flow. Compromised blood supply can explain the potential of non-union and avascular necrosis of the proximal pole. The healing process can be complicated by volar angulation of the fracture leading to humpback deformity. This will disrupt carpal kinematics, and result in lunate instability and dorsal intercalated segment instability (DISI). Untreated scaphoid non-union can lead to degenerative changes, called scaphoid non-union advanced collapse (SNAC), and irreversible impairment such as pain and altered hand function.

X-ray is commonly applied to evaluate the scaphoid, although CT scans are reportedly superior in terms of displacement, angulation and union[9]. Different measurements to describe the angulation and deformity of the scaphoid are suggested. The Height length ratio (HLR) and dorsal cortical angle (DCA) are found to be the most reliable measurements.

Surgical treatment of scaphoid delayed/non-union is technically demanding and often results in a long period with a supportive bandage until union is established. Current treatment strategies for delayed union and non-union include vascularized or non-vascularized bone graft with internal fixation. Kirchner wires or screws have been the gold standard for fixation.

Arthroscopic reconstruction with C chips and internal fixation is predominantly applied in delayed union and stable non-union. The advantages of arthroscopy include thorough wrist assessment, evaluation of concomitant ligamentous injury and minimal trauma to the ligament structures, joint capsule, and the tenuous blood supply.

The objective of this study protocol is to describe the methodology for a RCT comparing time to union and functional outcome scores of arthroscopic assisted C chips reconstruction or open C graft reconstruction for scaphoid delayed/non-union

Hypothesis:

Arthroscopic assisted C chips graft reconstruction of scaphoid delayed/non-union is superior to open C graft reconstruction regarding faster time to union, by at least mean 3 weeks difference.

Study design:

This is a single-center, 1:1 observer-blinded randomized controlled, superiority trial. The main objective is to compare open C graft with arthroscopic assisted C chips graft reconstruction for scaphoid fractures with delayed/non-union.

Subjects:

A total of 88 patients with scaphoid delayed/non-union are randomized to either:

1. Group A - Arthroscopic assisted C chips graft reconstruction (intervention group), n=44
2. Group O - Open C graft reconstruction (control group), n=44

Inclusion criteria:

1. Patients aged 18-68 years.
2. A scaphoid fracture without healing 2-6 months since fracture (delayed union) for cases with either displacement >1mm or comminution and failed non-operative treatment.
3. Scaphoid fracture without healing >6 months since fracture (non-union) regardless of displacement, comminution and if previous non-operative treatment has been tried.
4. ASA 1-3.

Exclusion criteria:

1. Open fractures
2. Associated trans-scaphoid perilunate dislocation.
3. Associated fracture in the hand/upper extremity.
4. Previous failed surgical treatment for scaphoid delayed/non-union.
5. Stage 2 SNAC or above.
6. Avascular necrosis of the proximal pole as evaluated with MRI and absence of punctate bleeding intraoperatively.
7. Patients with gross humpback deformity of HLR >0.75 and/or DCA <70⁰.
8. Patients unable to understand instructions in Danish, complete the rehabilitation protocol, or answering the questionnaires because of physical or cognitive impairment, as evaluated by the surgeon at the first visit.

Enrolment:

All Danish citizens aged 18-68 years with scaphoid delayed/non-union referred to the hand surgery unit, Herlev and Gentofte University Hospital, will be offered participation in the study. Other hand unit departments in the Capital Region of Denmark will forward their referrals to our department for inclusion. The physician will review the medical records and assess whether the patients fulfil the inclusion/exclusion criteria.

Patients will undergo a clinical examination and CT scan of the wrist to describe angulation (HLR and DCA), displacement, localization of non-union, presence of cysts, and degenerative changes. All patients with involvement of the proximal pole will undergo gadolinium-enhanced MRI to clarify vascularity, but the final assessment of avascular necrosis of the proximal pole will be performed perioperatively. If punctate bleeding after tourniquet being off for at least 5 minutes of expectation cannot be visible, the patient will then be excluded from the study and will be simultaneously operated with a vascular bone graft or a salvage procedure

Randomization:

Based on the sample size calculation, a total number of 88 patients will be allocated into two groups of equal size

1. Group A - Arthroscopic assisted C-chips graft reconstruction (intervention group), N=44.
2. Group O - Open C-only graft reconstruction (control group), N=44.

The randomization is done in the outpatient clinic and the patients will be informed about the operative treatment. The randomization application, Research Electronic Data Capture (REDCap), will allocate patients in a 1:1 ratio, stratified for proximal pole fracture (yes /no), dislocation (>/< 2mm), and smoking (yes/ no). A statistician will generate a randomization sequence for RED-Cap.

In this observer-blinded RCT, union is assessed by a blinded musculoskeletal radiologist. QDASH is a patient-reported survey, without the involvement of surgeons or research staff. Other secondary outcomes will be measured by an independent observer. The study will not be blinded to the operating theatre staff, surgeons, physiotherapists, or patients.

Clinical outcomes and patient-reported outcomes will be measured after 1.5, 3, 6, 12, and 24 months. Online questionnaires will be sent after 5 and 10 years.

Primary outcome is time to union, assessed with repeated CT-scans in two weeks interval from 6-16 weeks after operative treatment. Union will be proclaimed and recorded when >50% bone bridging occurs on CT.

Secondary outcomes are: Q-DASH (patient reported outcome, questionnaire), range of Motion, grip strength and Key pinch (functional outcome). Finally, pain and donor site morbidity evaluated with VAS, Complications, EQ5D-5L (cost-utility measure) and patient satisfaction are recorded.

The study will follow the Helsinki Declaration. All patients will receive oral and written information before the assignment of consent. Patients can withdraw their consent at any time. The Danish National Committee on Health Research Ethics has approved this study protocol (Journal-nr.: H-21075664). All patients in the study are covered by the insurance policies of ordinary treatment regarding complaints and compensation following the rules in the Act on Complaints and Compensation in the Health Services in Denmark.

The background radiation in Denmark is 3 mSv pr. Year. The radiation dosage due to repeated CT scans of 0.03mSv, is a maximum 0.21mSv corresponding to approximately 21 days of background radiation.

Patients with prolonged period to union or failed union are at risk of the increased radiation dosage compared to case/surgeon-specific conditions as standard treatment. The current standard treatment at our department includes follow up until the union is established. In this study, we will have additional follow-up examinations at 6 months and at 1 and 2 years. It has the risk of keeping the patients in the role of being ill. However, the patients can have a feeling of extra good care with the possibility to address uncertainty or problems more easily.

Patients are at risk of being treated inferior with an intervention which is deemed inferior with the study analysis, but nothing a priori suggests which intervention is the better one.

The trial will provide high-quality evidence regarding time to union, short- and long-term functional outcomes of open and arthroscopic assisted graft reconstruction for scaphoid delayed/non-union.

The results from the study can contribute to establish a treatment algorithm for scaphoid delayed/non-union together with results from other studies.

Neither the primary investigator, participation investigators, and sponsors have personal economic interests in the results of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-68 years.
2. A scaphoid fracture without healing 2-6 months since fracture (delayed union) for cases with either displacement >1mm or comminution and failed non-operative treatment.
3. Scaphoid fracture without healing >6 months since fracture (non-union) regardless of displacement, comminution and if previous non-operative treatment has been tried.
4. ASA 1-3.

Exclusion Criteria:

1. Open fractures
2. Associated trans-scaphoid perilunate dislocation.
3. Associated fracture in the hand/upper extremity.
4. Previous failed surgical treatment for scaphoid delayed/non-union.
5. Stage 2 SNAC or above.
6. Avascular necrosis of the proximal pole as evaluated with MRI and absence of punctate bleeding intraoperatively.
7. Patients with gross humpback deformity of HLR >0.75 and/or DCA <70⁰.
8. Patients unable to understand instructions in Danish, complete the rehabilitation protocol, or answering the questionnaires because of physical or cognitive impairment, as evaluated by the surgeon at the first visit.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to Union | 6-16 weeks postoperative in 2 weeks intervals. If unions is not achieved a CT will be made 26 weeks postoperatively. If union is not achieved at that point, the patient will be presented for another treatment modality
  Assessed with CT-scans. Union is proclaimed if at least 50% bone bridging is recorded together with absence of pain in the clinical examination

SECONDARY OUTCOMES:
The Quick Disability of the Arm, Shoulder, and Hand (Q-DASH) | Preoperatively, 1.5 md, 3md, 6md, 12md, 24md, 60md, and 120 months postoperative
  Q Dash is a patient-reported survey. It is a subset of 11 items from the 30-item DASH questions that assess difficulties with specific tasks: 5 concerning symptoms, 4 on social function, and 1 on work function, sleep, and confidence. The score ranges from 0-100 and the higher score reflects disabilities. The MCID has been defined as 10.8 (range, 5-15) for comparable patients.
Union rate | 6-16 weeks postoperative. If unions is not achieved a CT will be made 26 weeks postoperatively
  Assessed with CT-scans
Correction of deformity | Before surgery compared to CT-scan with >50% bone bridging.
  The Height length ratio (HLR) and dorsal cortical angle (DCA) are found to be the most reliable measurements to describe angulation. The height-length ratio is calculated by dividing the scaphoid height by length.
Pain (VAS) | Preoperatively, 1.5, 3, 6, 12, 24, 60, and 120 months postoperative
  Pain at rest and activity is recorded on a visual analogue scale (VAS), ranging from 0-10, with 10 reflecting the worst and 0 representing no pain in the wrist.
Donor site morbidity | Preoperatively, 1.5, 3, 6, 12, 24, 60, and 120 months postoperative
  located to the iliac crest (Group O) and distal radius (Group A) are evaluated with VAS ranging from 0-10, with 10 reflecting the worst and 0 representing no pain in the wrist
Grip strength | Preoperatively, 1.5, 3, 6, 12, and 24 months postoperative
  is measured in kilograms with a Jamar dynamometer with the elbow will be in 90° flexion and attached to the chest compared to the unaffected.
Key pinch | Preoperatively, 1.5, 3, 6, 12, 24, 60, and 120 months postoperative
  is measured in kilograms using a pinch gauge with the elbow in in 90° flexion and attached to the chest, compared to the unaffected wrist.

OTHER OUTCOMES:
Patient satisfaction | Preoperatively, 1.5, 3, 6, 12, 24, 60, and 120 months postoperative
  is evaluated with the following question: What is the function of your hand today, compared to before surgery? With the following answer options: (1) disaster, (2) much worse, (3) slightly worse, (4) unchanged, (5) slightly better, (6) much better, (7) recovered. Secondary, for future research perspective patients are asked: When you consider the following parameters: The activities you can carry out in daily life, your pain, your function of the hand, do you think your current situation is satisfactory? (yes/no).
EQ5D-5L | Baseline and 2-year follow up scores will be compared
  will be used to estimate the threshold for acceptable cost-utility ratio - the threshold for how much health care providers will pay for an extra quality-adjusted life year (QALY). The cost utility of the Arthroscopic- and open technique will be compared. A cost model will be defined from patient data, clinical records, and unit costs from the Danish health care system. Length of hospital stay, discharge, pain medication usage and readmission will be recorded.
Complications and secondary surgery | Preoperatively, 1.5, 3, 6, 12 and 24 months postoperative
  We will record all complications related to the operative treatment (Tendon-, ligament-, nerve- or arterial injury, infection, complex regional pain syndrome, hematoma, or hardware failure). Reoperations, defined as revision surgery and secondary surgery due to no union will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gvozdenoviz, MD, Principal Investigator — Orthopedic department, Copenhagen university hospital Gentofte Hospital
Locations (1):
- University Hospital Herlev/Gentofte, Department of Orthopedic Surgery, Clinic for Shoulder-, Elbow- and Hand Surgery, Hellerup, Denmark, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The dataset and results will be available from the primary investigator on request, with acceptance of the the Danish Data Protection Agency (Pactius).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available when the study results are published. The data will be available for 10 years after finishing of recruitment, as accepted by the Danish Data Protection Agency (Pactius).
Access Criteria: On request with relevant argumentation for intended use, and acceptance by the data protection agency.

REFERENCES:
- [Background] Jorgsholm P, Ossowski D, Thomsen N, Bjorkman A. Epidemiology of scaphoid fractures and non-unions: A systematic review. Handchir Mikrochir Plast Chir. 2020 Sep;52(5):374-381. doi: 10.1055/a-1250-8190. Epub 2020 Sep 29. PMID 32992390
- [Background] Cooney WP 3rd, Dobyns JH, Linscheid RL. Nonunion of the scaphoid: analysis of the results from bone grafting. J Hand Surg Am. 1980 Jul;5(4):343-54. doi: 10.1016/s0363-5023(80)80173-0. PMID 6999072
- [Background] Linscheid RL, Dobyns JH, Beabout JW, Bryan RS. Traumatic instability of the wrist: diagnosis, classification, and pathomechanics. J Bone Joint Surg Am. 2002 Jan;84(1):142. doi: 10.2106/00004623-200201000-00020. No abstract available. PMID 11792792
- [Background] Grewal R, Suh N, MacDermid JC. The Missed Scaphoid Fracture-Outcomes of Delayed Cast Treatment. J Wrist Surg. 2015 Nov;4(4):278-83. doi: 10.1055/s-0035-1564983. PMID 26649260
- [Background] Little CP, Burston BJ, Hopkinson-Woolley J, Burge P. Failure of surgery for scaphoid non-union is associated with smoking. J Hand Surg Br. 2006 Jun;31(3):252-5. doi: 10.1016/j.jhsb.2005.12.010. Epub 2006 Feb 20. PMID 16488521
- [Background] Schuind F, Moungondo F, El Kazzi W. Prognostic factors in the treatment of carpal scaphoid non-unions. Eur J Orthop Surg Traumatol. 2017 Jan;27(1):3-9. doi: 10.1007/s00590-016-1886-4. Epub 2016 Nov 28. PMID 27896458
- [Background] Grewal R, Suh N, Macdermid JC. Use of computed tomography to predict union and time to union in acute scaphoid fractures treated nonoperatively. J Hand Surg Am. 2013 May;38(5):872-7. doi: 10.1016/j.jhsa.2013.01.032. Epub 2013 Mar 23. PMID 23531510
- [Background] Ramamurthy C, Cutler L, Nuttall D, Simison AJ, Trail IA, Stanley JK. The factors affecting outcome after non-vascular bone grafting and internal fixation for nonunion of the scaphoid. J Bone Joint Surg Br. 2007 May;89(5):627-32. doi: 10.1302/0301-620X.89B5.18183. PMID 17540748
- [Background] Buijze GA, Wijffels MM, Guitton TG, Grewal R, van Dijk CN, Ring D; Science of Variation Group. Interobserver reliability of computed tomography to diagnose scaphoid waist fracture union. J Hand Surg Am. 2012 Feb;37(2):250-4. doi: 10.1016/j.jhsa.2011.10.051. PMID 22281168
- [Background] Guldbrandsen CW, Radev DI, Gvozdenovic R. Normal ranges for measurements of the scaphoid bone from sagittal computed tomography images. J Hand Surg Eur Vol. 2021 Jul;46(6):594-599. doi: 10.1177/1753193420987522. Epub 2021 Jan 17. PMID 33459143
- [Background] Bain GI, Bennett JD, MacDermid JC, Slethaug GP, Richards RS, Roth JH. Measurement of the scaphoid humpback deformity using longitudinal computed tomography: intra- and interobserver variability using various measurement techniques. J Hand Surg Am. 1998 Jan;23(1):76-81. doi: 10.1016/S0363-5023(98)80093-2. PMID 9523959
- [Background] Merrell GA, Wolfe SW, Slade JF 3rd. Treatment of scaphoid nonunions: quantitative meta-analysis of the literature. J Hand Surg Am. 2002 Jul;27(4):685-91. doi: 10.1053/jhsu.2002.34372. PMID 12132096
- [Background] Sayegh ET, Strauch RJ. Graft choice in the management of unstable scaphoid nonunion: a systematic review. J Hand Surg Am. 2014 Aug;39(8):1500-6.e7. doi: 10.1016/j.jhsa.2014.05.009. Epub 2014 Jul 3. PMID 24997785
- [Background] Huang YC, Liu Y, Chen TH. Long-term results of scaphoid nonunion treated by intercalated bone grafting and Herbert's screw fixation--a study of 49 patients for at least five years. Int Orthop. 2009 Oct;33(5):1295-300. doi: 10.1007/s00264-008-0663-3. Epub 2008 Oct 28. PMID 18956188
- [Background] Goyal T, Sankineani SR, Tripathy SK. Local distal radius bone graft versus iliac crest bone graft for scaphoid nonunion: a comparative study. Musculoskelet Surg. 2013 Aug;97(2):109-14. doi: 10.1007/s12306-012-0219-y. Epub 2012 Sep 12. PMID 22968662
- [Background] Oh WT, Kang HJ, Chun YM, Koh IH, Lee YJ, Choi YR. Retrospective Comparative Outcomes Analysis of Arthroscopic Versus Open Bone Graft and Fixation for Unstable Scaphoid Nonunions. Arthroscopy. 2018 Oct;34(10):2810-2818. doi: 10.1016/j.arthro.2018.04.024. Epub 2018 Aug 30. PMID 30173911
- [Background] Chu PJ, Shih JT. Arthroscopically assisted use of injectable bone graft substitutes for management of scaphoid nonunions. Arthroscopy. 2011 Jan;27(1):31-7. doi: 10.1016/j.arthro.2010.05.015. Epub 2010 Oct 8. PMID 20934844
- [Background] Lee YK, Choi KW, Woo SH, Ho PC, Lee M. The clinical result of arthroscopic bone grafting and percutaneous K-wires fixation for management of scaphoid nonunions. Medicine (Baltimore). 2018 Mar;97(13):e9987. doi: 10.1097/MD.0000000000009987. PMID 29595703
- [Background] Slade JF 3rd, Geissler WB, Gutow AP, Merrell GA. Percutaneous internal fixation of selected scaphoid nonunions with an arthroscopically assisted dorsal approach. J Bone Joint Surg Am. 2003;85-A Suppl 4:20-32. doi: 10.2106/00004623-200300004-00003. PMID 14652390
- [Background] Kim JP, Seo JB, Yoo JY, Lee JY. Arthroscopic management of chronic unstable scaphoid nonunions: effects on restoration of carpal alignment and recovery of wrist function. Arthroscopy. 2015 Mar;31(3):460-9. doi: 10.1016/j.arthro.2014.08.035. Epub 2014 Nov 4. PMID 25442643
- [Background] Kang HJ, Chun YM, Koh IH, Park JH, Choi YR. Is Arthroscopic Bone Graft and Fixation for Scaphoid Nonunions Effective? Clin Orthop Relat Res. 2016 Jan;474(1):204-12. doi: 10.1007/s11999-015-4495-3. Epub 2015 Aug 7. PMID 26250139
- [Background] Cognet JM, Louis P, Martinache X, Schernberg F. Arthroscopic grafting of scaphoid nonunion - surgical technique and preliminary findings from 23 cases. Hand Surg Rehabil. 2017 Feb;36(1):17-23. doi: 10.1016/j.hansur.2016.11.002. Epub 2016 Dec 29. PMID 28137436
- [Background] Hsiung W, Huang HK, Wang JP, Chang MC, Huang YC. Arthroscopic realignment and osteosynthesis of unstable scaphoid nonunion with cancellous bone graft from the ipsilateral radius. Int Orthop. 2021 Jan;45(1):191-197. doi: 10.1007/s00264-020-04840-2. Epub 2020 Oct 13. PMID 33048201
- [Background] Waitayawinyu T, Lertcheewanan W, Boonyasirikool C, Niempoog S. Arthroscopic Treatment of Scaphoid Nonunion With Olecranon Bone Graft and Screw Fixation Leads to Union and Improved Outcomes. Arthroscopy. 2022 Mar;38(3):761-772. doi: 10.1016/j.arthro.2021.09.018. Epub 2021 Sep 25. PMID 34571185
- [Background] Hackney LA, Dodds SD. Assessment of scaphoid fracture healing. Curr Rev Musculoskelet Med. 2011 Mar 8;4(1):16-22. doi: 10.1007/s12178-011-9072-0. PMID 21475561
- [Background] Hannemann PF, Brouwers L, van der Zee D, Stadler A, Gottgens KW, Weijers R, Poeze M, Brink PR. Multiplanar reconstruction computed tomography for diagnosis of scaphoid waist fracture union: a prospective cohort analysis of accuracy and precision. Skeletal Radiol. 2013 Oct;42(10):1377-82. doi: 10.1007/s00256-013-1658-8. Epub 2013 Jun 6. PMID 23740357
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Gummesson C, Ward MM, Atroshi I. The shortened disabilities of the arm, shoulder and hand questionnaire (QuickDASH): validity and reliability based on responses within the full-length DASH. BMC Musculoskelet Disord. 2006 May 18;7:44. doi: 10.1186/1471-2474-7-44. PMID 16709254
- [Background] Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther. 2014 Jan;44(1):30-9. doi: 10.2519/jospt.2014.4893. Epub 2013 Oct 30. PMID 24175606
- [Background] Roh YH, Noh JH, Lee BK, Baek JR, Oh JH, Gong HS, Baek GH. Reliability and validity of carpal alignment measurements in evaluating deformities of scaphoid fractures. Arch Orthop Trauma Surg. 2014 Jun;134(6):887-93. doi: 10.1007/s00402-014-1998-4. Epub 2014 Apr 23. PMID 24756533
- [Background] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Background] Mathiowetz V, Weber K, Volland G, Kashman N. Reliability and validity of grip and pinch strength evaluations. J Hand Surg Am. 1984 Mar;9(2):222-6. doi: 10.1016/s0363-5023(84)80146-x. PMID 6715829
- [Background] Kvien TK, Heiberg T, Hagen KB. Minimal clinically important improvement/difference (MCII/MCID) and patient acceptable symptom state (PASS): what do these concepts mean? Ann Rheum Dis. 2007 Nov;66 Suppl 3(Suppl 3):iii40-1. doi: 10.1136/ard.2007.079798. PMID 17934093
- [Background] Pinder RM, Brkljac M, Rix L, Muir L, Brewster M. Treatment of Scaphoid Nonunion: A Systematic Review of the Existing Evidence. J Hand Surg Am. 2015 Sep;40(9):1797-1805.e3. doi: 10.1016/j.jhsa.2015.05.003. Epub 2015 Jun 24. PMID 26116095
- [Background] Hegazy G, Massoud AH, Seddik M, Abd-Elghany T, Abdelaal M, Saqr Y, Abdelaziz M, Zayed E, Hassan M. Structural Versus Nonstructural Bone Grafting for the Treatment of Unstable Scaphoid Waist Nonunion Without Avascular Necrosis: A Randomized Clinical Trial. J Hand Surg Am. 2021 Jun;46(6):462-470. doi: 10.1016/j.jhsa.2021.01.027. Epub 2021 Apr 1. PMID 33814250
- [Background] Kim JK, Yoon JO, Baek H. Corticocancellous bone graft vs cancellous bone graft for the management of unstable scaphoid nonunion. Orthop Traumatol Surg Res. 2018 Feb;104(1):115-120. doi: 10.1016/j.otsr.2017.11.011. Epub 2017 Dec 16. PMID 29258960
- [Background] Cohen MS, Jupiter JB, Fallahi K, Shukla SK. Scaphoid waist nonunion with humpback deformity treated without structural bone graft. J Hand Surg Am. 2013 Apr;38(4):701-5. doi: 10.1016/j.jhsa.2012.12.030. Epub 2013 Feb 13. PMID 23415167
- [Background] Yang H, Bullock WA, Myhal A, DeShield P, Duffy D, Main RP. Cancellous Bone May Have a Greater Adaptive Strain Threshold Than Cortical Bone. JBMR Plus. 2021 Mar 30;5(5):e10489. doi: 10.1002/jbm4.10489. eCollection 2021 May. PMID 33977205
- [Background] Singh HP, Forward D, Davis TR, Dawson JS, Oni JA, Downing ND. Partial union of acute scaphoid fractures. J Hand Surg Br. 2005 Oct;30(5):440-5. doi: 10.1016/j.jhsb.2005.05.007. PMID 16006021
- [Background] Lozano-Calderon S, Blazar P, Zurakowski D, Lee SG, Ring D. Diagnosis of scaphoid fracture displacement with radiography and computed tomography. J Bone Joint Surg Am. 2006 Dec;88(12):2695-703. doi: 10.2106/JBJS.E.01211. PMID 17142420
- [Background] Dias JJ, Taylor M, Thompson J, Brenkel IJ, Gregg PJ. Radiographic signs of union of scaphoid fractures. An analysis of inter-observer agreement and reproducibility. J Bone Joint Surg Br. 1988 Mar;70(2):299-301. doi: 10.1302/0301-620X.70B2.3346310.
- [Background] Hannemann PFW, Brouwers L, Dullaert K, van der Linden ES, Poeze M, Brink PRG. Determining scaphoid waist fracture union by conventional radiographic examination: an analysis of reliability and validity. Arch Orthop Trauma Surg. 2015 Feb;135(2):291-296. doi: 10.1007/s00402-014-2147-9. Epub 2015 Jan 3. PMID 25555379
- [Background] Farracho LC, Moutinot B, Neroladaki A, Hamard M, Gorican K, Poletti PA, Beaulieu JY, Bouvet C, Boudabbous S. Determining diagnosis of scaphoid healing: Comparison of cone beam CT and X-ray after six weeks of immobilization. Eur J Radiol Open. 2020 Sep 2;7:100251. doi: 10.1016/j.ejro.2020.100251. eCollection 2020. PMID 32944592
- [Background] Biswas D, Bible JE, Bohan M, Simpson AK, Whang PG, Grauer JN. Radiation exposure from musculoskeletal computerized tomographic scans. J Bone Joint Surg Am. 2009 Aug;91(8):1882-9. doi: 10.2106/JBJS.H.01199. PMID 19651945
- [Background] Zhou Q. [Recommendations for the conduct, reporting, editing and publication of scholarly work in medical journals]. Zhonghua Gan Zang Bing Za Zhi. 2014 Oct;22(10):781-91. No abstract available. Chinese. PMID 25558501
- [Background] World Medical Association Inc. Declaration of Helsinki. Ethical principles for medical research involving human subjects. J Indian Med Assoc. 2009 Jun;107(6):403-5. No abstract available. PMID 19886379
- [Derived] Kjaer M, Rasmussen JV, Gvozdenovic R. Arthroscopic versus open cancellous bone grafting for scaphoid delayed/nonunion in adults (SCOPE-OUT): study protocol for a randomized clinical trial. Trials. 2023 Apr 14;24(1):273. doi: 10.1186/s13063-023-07281-5. PMID 37060040